CLINICAL TRIAL: NCT00641043
Title: A Randomised, Double-blind, Placebo Controlled, Parallel Group 24 Week Study to Assess the Efficacy and Safety of BI 1356 (5 mg) in Combination With 30 mg Pioglitazone (Both Administered Orally Once Daily), Compared to 30 mg Pioglitazone Plus Placebo in Drug Naive or Previously Treated Type 2 Diabetic Patients With Insufficient Glycaemic Control.
Brief Title: Efficacy vs Placebo as Initial Combination Therapy With Pioglitazone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1218.15; 2007-002456-41 (EudraCT Number: EudraCT)
Record Dates: First submitted 2008-02-29; First posted 2008-03-21 (Estimated); Results first posted 2011-06-07 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone; Linagliptin

ARMS (2):
- BI 1356 (5 mg) (Experimental): BI 1356 5mg in initial combination therapy with pioglitazone 30 mg
  Interventions: Drug: Linagliptin + pioglitazone (30 mg)
- Placebo matching BI 1356 5 mg (Placebo Comparator): Placebo in initial combination therapy with pioglitazone 30 mg
  Interventions: Drug: placebo + pioglitazone (30 mg)

INTERVENTIONS:
Drug: placebo + pioglitazone (30 mg) — placebo + overcapsulated 30 mg tablet, once daily
  Arms: Placebo matching BI 1356 5 mg
Drug: Linagliptin + pioglitazone (30 mg) — 5 mg tablet + overcapsulated 30 mg tablet, once daily
  Arms: BI 1356 (5 mg)

SUMMARY:
The objective of the current study is to investigate the efficacy, safety and tolerability of BI 1356 (Linagliptin) (5 mg / once daily) compared to placebo given for 24 weeks as initial combination therapy with pioglitazone 30 mg in patients with type 2 diabetes mellitus with insufficient glycaemic control.

ELIGIBILITY:
Inclusion criteria:

1. Signed and dated written Informed Consent (IC) by date of Visit 1a in accordance with Good Clinical Practice (GCP) and local legislation
2. Patients with a diagnosis of type 2 diabetes mellitus and treatment naive or previously treated with any oral hypoglycaemic agent; antidiabetic therapy has to be unchanged for ten weeks prior to informed consent.
3. Glycosylated haemoglobin A1 (HbA1c) 7.5-11% at Visit 2 (Start of Run-in).
4. Male and female patients aged > or = 18 and < or = to 80 years at Visit 1a (Screening).
5. Body Mass Index (BMI) < or = 40 kg/m2 at Visit 1a (Screening)
6. Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation.

Exclusion criteria:

1. Myocardial infarction, stroke or Transient Isquemic Atack (TIA) within 6 months prior to Inform Consent (IC)
2. Impaired hepatic function, defined by serum levels of either Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), or alkaline phosphatase above 3 x upper limit of normal (ULN) determined at Visit 1a.
3. Known hypersensitivity or allergy to the investigational product or its excipients and/or to hydrochloride of pioglitazone or its excipients
4. Treatment with Glucagon-like peptide-1 (GLP-1) analogue / agonist within 3 months prior to IC.
5. Treatment with insulin within 3 months prior to IC
6. Treatment with anti-obesity drugs 3 months prior to IC.
7. Alcohol abuse within the 3 months prior to IC that would interfere with trial participation or drug abuse.
8. Participation in another trial with an investigational drug within 2 months prior to IC.
9. Fasting blood glucose > 240 mg/dl (=13.3 mmol/L) at screening (Visit 1).
10. Pre-menopausal women (last menstruation < or =1 year prior to signing IC) who:

    * are nursing or pregnant,
    * or are of child-bearing potential and are not practicing an acceptable method of birth control, or do not plan to continue using this method throughout the study and do not agree to submit to periodic pregnancy testing during participation in the trial. Acceptable methods of birth control include transdermal patch, intra uterine devices/systems (IUDs/IUSs), oral, implantable or injectable contraceptives, sexual abstinence and vasectomised partner. No exception will be made.
11. Treatment with systemic steroids or change in the dosage of thyroid hormone within six weeks prior to IC
12. Heart failure New York Heart Asociation (NYHA) class I-IV, or history of heart failure.
13. Diabetic ketoacidosis within 6 months prior to IC.
14. Hemodialyzed patients due to limited experience with Thiazolidinediones (TZDs)
15. Any other clinical condition wich, in the opinion of the investigator, would not alow safe completion of the protocol and safe administration of BI1356 and pioglitazone.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2008-03; Primary Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (43):
- Austria (4):
  - 1218.15.43004 Boehringer Ingelheim Investigational Site, Feldkirch
  - 1218.15.43001 Boehringer Ingelheim Investigational Site, Graz
  - 1218.15.43003 Boehringer Ingelheim Investigational Site, Vienna
  - 1218.15.43005 Boehringer Ingelheim Investigational Site, Vienna
- Greece (8):
  - 1218.15.30004 Boehringer Ingelheim Investigational Site, Athens
  - 1218.15.30007 Boehringer Ingelheim Investigational Site, Athens
  - 1218.15.30017 Boehringer Ingelheim Investigational Site, Ioannina
  - 1218.15.30002 Boehringer Ingelheim Investigational Site, Melissia-Athens
  - 1218.15.30003 Boehringer Ingelheim Investigational Site, Nikaia
  - 1218.15.30006 Boehringer Ingelheim Investigational Site, Thessaloniki
  - 1218.15.30014 Boehringer Ingelheim Investigational Site, Thessaloniki
  - 1218.15.30016 Boehringer Ingelheim Investigational Site, Thessaloniki
- Hungary (6):
  - 1218.15.36003 Boehringer Ingelheim Investigational Site, Budapest
  - 1218.15.36004 Boehringer Ingelheim Investigational Site, Budapest
  - 1218.15.36006 Boehringer Ingelheim Investigational Site, Budapest
  - 1218.15.36008 Boehringer Ingelheim Investigational Site, Debrecen
  - 1218.15.36005 Boehringer Ingelheim Investigational Site, Győr
  - 1218.15.36002 Boehringer Ingelheim Investigational Site, Szombathely
- Japan (5):
  - 1218.15.81001 Boehringer Ingelheim Investigational Site, Amagasaki, Hyogo
  - 1218.15.81005 Boehringer Ingelheim Investigational Site, Koganei, Tokyo
  - 1218.15.81002 Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - 1218.15.81004 Boehringer Ingelheim Investigational Site, Shinjyuku-ku,Tokyo
  - 1218.15.81003 Boehringer Ingelheim Investigational Site, Suita, Osaka,
- Portugal (2):
  - 1218.15.35007 Boehringer Ingelheim Investigational Site, Aveiro
  - 1218.15.35001 Boehringer Ingelheim Investigational Site, Lisbon
- Romania (5):
  - 1218.15.40504 Boehringer Ingelheim Investigational Site, Alba Iulia
  - 1218.15.40501 Boehringer Ingelheim Investigational Site, Bucharest
  - 1218.15.40502 Boehringer Ingelheim Investigational Site, Bucharest
  - 1218.15.40503 Boehringer Ingelheim Investigational Site, Sibiu
  - 1218.15.40505 Boehringer Ingelheim Investigational Site, Târgu Mureş
- Spain (13):
  - 1218.15.34002 Boehringer Ingelheim Investigational Site, Badalona
  - 1218.15.34011 Boehringer Ingelheim Investigational Site, Badia Del Vallés
  - 1218.15.34001 Boehringer Ingelheim Investigational Site, Bercelona
  - 1218.15.34012 Boehringer Ingelheim Investigational Site, Borges Del Camp
  - 1218.15.34013 Boehringer Ingelheim Investigational Site, Centelles
  - 1218.15.34007 Boehringer Ingelheim Investigational Site, Granada
  - 1218.15.34008 Boehringer Ingelheim Investigational Site, L'Hospitalet de Llobregat (Barcelona)
  - 1218.15.34009 Boehringer Ingelheim Investigational Site, L'Hospitalet de Llobregat (Barcelona)
  - 1218.15.34004 Boehringer Ingelheim Investigational Site, Madrid
  - 1218.15.34006 Boehringer Ingelheim Investigational Site, Madrid
  - 1218.15.34010 Boehringer Ingelheim Investigational Site, Sant Adrià Del Besós (Barcelona)
  - 1218.15.34005 Boehringer Ingelheim Investigational Site, Seville
  - 1218.15.34014 Boehringer Ingelheim Investigational Site, Vic (Barcelona)

REFERENCES:
- [Derived] Johansen OE, Neubacher D, von Eynatten M, Patel S, Woerle HJ. Cardiovascular safety with linagliptin in patients with type 2 diabetes mellitus: a pre-specified, prospective, and adjudicated meta-analysis of a phase 3 programme. Cardiovasc Diabetol. 2012 Jan 10;11:3. doi: 10.1186/1475-2840-11-3. PMID 22234149

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo + Pioglitazone: Patients randomized to receive treatment with matching placebo (to Linagliptin 5 mg) and Pioglitazone 30 mg
- Linagliptin + Pioglitazone: Patients randomized to receive treatment with Linagliptin 5 mg and Pioglitazone 30 mg
Period: Overall Study
Arm/Group | Placebo + Pioglitazone | Linagliptin + Pioglitazone
Started | 130 (number who started treatment) | 259 (number who started treatment)
Completed | 111 (number who completed treatment) | 244 (number who completed treatment)
Not Completed | 19 | 15
Not completed — Adverse Event | 6 | 4
Not completed — Protocol Violation | 2 | 3
Not completed — Lost to Follow-up | 3 | 2
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Other incl. lack of efficacy | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Pioglitazone | Linagliptin + Pioglitazone | Total
Number analyzed (Participants) | 130 | 259 | 389
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.1 (10.1) | 57.7 (9.6) | 57.5 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 107 | 152
  Male | 85 | 152 | 237
Body mass index continuous [Mean (Standard Deviation); unit: kg/m^2] | 29.72 (4.84) | 28.68 (4.82) | 29.02 (4.85)
Glycosylated haemoglobin A1 (HbA1c) [Mean (Standard Deviation); unit: Percent] | 8.58 (0.87) | 8.60 (0.79) | 8.59 (0.82)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] | 190.3 (43.8) | 189.8 (42.7) | 189.9 (43.0)

OUTCOME MEASURES:

1. Primary Outcome: HbA1c Change From Baseline to Week 24
Description: HbA1c is measured as a percentage. Thus, this change from baseline reflects the Week 24 HbA1c percent minus the baseline HbA1c percent. Means are treatment adjusted for baseline HbA1c and previous anti-diabetic medication.
Time Frame: Baseline and week 24
Population: The Full Analysis Set (FAS) included all treated and randomised patients with a baseline and at least one on treatment HbA1c measurement available. Last observation carried forward (LOCF) was used as the imputation rule.
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Placebo + Pioglitazone | Linagliptin + Pioglitazone
Number analyzed (Participants) | 128 | 252
Percent | -0.56 (0.09) | -1.06 (0.06)
Statistical Analysis 1: Comparison: Placebo + Pioglitazone vs Linagliptin + Pioglitazone; Linagliptin vs. Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.51, 95% CI [-0.71 to -0.30], Standard Error of Mean 0.10

2. Secondary Outcome: HbA1c Change From Baseline to Week 6
Description: HbA1c is measured as a percentage. Thus, this change from baseline reflects the Week 6 HbA1c percent minus the baseline HbA1c percent. Means are treatment adjusted for baseline HbA1c and previous anti-diabetic medication.
Time Frame: Baseline and week 6
Population: The Full Analysis Set (FAS) included all randomised and treated patients with a baseline and at least one on treatment HbA1c measurement available. Last observation carried forward (LOCF) was used as the imputation rule.
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Placebo + Pioglitazone | Linagliptin + Pioglitazone
Number analyzed (Participants) | 128 | 252
Percent | -0.03 (0.06) | -0.41 (0.04)
Statistical Analysis 1: Comparison: Placebo + Pioglitazone vs Linagliptin + Pioglitazone; Linagliptin vs. Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.38, 95% CI [-0.52 to -0.24], Standard Error of Mean 0.07

3. Secondary Outcome: HbA1c Change From Baseline to Week 12
Description: HbA1c is measured as a percentage. Thus, this change from baseline reflects the Week 12 HbA1c percent minus the baseline HbA1c percent. Means are treatment adjusted for baseline HbA1c and previous anti-diabetic medication.
Time Frame: Baseline and week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Placebo + Pioglitazone | Linagliptin + Pioglitazone
Number analyzed (Participants) | 128 | 252
Percent | -0.35 (0.07) | -0.85 (0.05)
Statistical Analysis 1: Comparison: Placebo + Pioglitazone vs Linagliptin + Pioglitazone; Linagliptin vs. Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.50, 95% CI [-0.67 to -0.32], Standard Error of Mean 0.09

4. Secondary Outcome: HbA1c Change From Baseline to Week 18
Description: HbA1c is measured as a percentage. Thus, this change from baseline reflects the Week 18 HbA1c percent minus the baseline HbA1c percent. Means are treatment adjusted for baseline HbA1c and previous anti-diabetic medication.
Time Frame: Baseline and week 18
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Placebo + Pioglitazone | Linagliptin + Pioglitazone
Number analyzed (Participants) | 128 | 252
Percent | -0.55 (0.08) | -1.06 (0.06)
Statistical Analysis 1: Comparison: Placebo + Pioglitazone vs Linagliptin + Pioglitazone; Linagliptin vs. Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.51, 95% CI [-0.70 to -0.32], Standard Error of Mean 0.10

5. Secondary Outcome: FPG Change From Baseline to Week 24
Description: This change from baseline reflects the Week 24 FPG minus the baseline FPG. Means are treatment adjusted for baseline HbA1c, baseline FPG and previous anti-diabetic medication.
Time Frame: Baseline and week 24
Population: This population includes the FAS using the LOCF imputation, with the further restriction of patients with a baseline and post-baseline FPG value.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo + Pioglitazone | Linagliptin + Pioglitazone
Number analyzed (Participants) | 122 | 243
mg/dL | -18.4 (3.0) | -32.6 (2.2)
Statistical Analysis 1: Comparison: Placebo + Pioglitazone vs Linagliptin + Pioglitazone; Linagliptin vs. Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -14.2, 95% CI [-21.1 to -7.3], Standard Error of Mean 3.5

6. Secondary Outcome: FPG Change From Baseline to Week 6
Description: This change from baseline reflects the Week 6 FPG minus the baseline FPG. Means are treatment adjusted for baseline HbA1c, baseline FPG and previous anti-diabetic medication.
Time Frame: Baseline and week 6
Population: as for outcome 5
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo + Pioglitazone | Linagliptin + Pioglitazone
Number analyzed (Participants) | 122 | 243
mg/dL | -17.0 (2.5) | -33.3 (1.9)
Statistical Analysis 1: Comparison: Placebo + Pioglitazone vs Linagliptin + Pioglitazone; Linagliptin vs. Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -16.4, 95% CI [-22.3 to -10.5], Standard Error of Mean 3.0

7. Secondary Outcome: FPG Change From Baseline to Week 12
Description: This change from baseline reflects the Week 12 FPG minus the baseline FPG. Means are treatment adjusted for baseline HbA1c, baseline FPG and previous anti-diabetic medication.
Time Frame: Baseline and week 12
Population: as for outcome 5
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo + Pioglitazone | Linagliptin + Pioglitazone
Number analyzed (Participants) | 122 | 243
mg/dL | -20.5 (2.7) | -33.8 (2.0)
Statistical Analysis 1: Comparison: Placebo + Pioglitazone vs Linagliptin + Pioglitazone; Linagliptin vs. Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -13.2, 95% CI [-19.5 to -7.0], Standard Error of Mean 3.2

8. Secondary Outcome: FPG Change From Baseline to Week 18
Description: This change from baseline reflects the Week 18 FPG minus the baseline FPG. Means are treatment adjusted for baseline HbA1c, baseline FPG and previous anti-diabetes medication.
Time Frame: Baseline and week 18
Population: as for outcome 5
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo + Pioglitazone | Linagliptin + Pioglitazone
Number analyzed (Participants) | 122 | 243
mg/dL | -19.3 (2.9) | -33.2 (2.1)
Statistical Analysis 1: Comparison: Placebo + Pioglitazone vs Linagliptin + Pioglitazone; Linagliptin vs. Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -13.9, 95% CI [-20.5 to -7.3], Standard Error of Mean 3.4

9. Secondary Outcome: Percentage of Patients With HbA1c <7.0% at Week 24
Description: The percentage of patients with an HbA1c value below 7% at week 24 was calculated for each treatment arm. If a patient did not have an HbA1c value at week 24 they were considered a failure, so HbA1c above 7%. Only patients with baseline HbA1c >= 7%
Time Frame: Baseline and Week 24
Population: This population includes the FAS with baseline HbA1c >= 7.0%. Non-completers were considered as failure imputation (NCF).
Measure: Number; unit: percentage of patients
Arm/Group | Placebo + Pioglitazone | Linagliptin + Pioglitazone
Number analyzed (Participants) | 128 | 252
percentage of patients | 30.5 (0) | 42.9 (0)
Statistical Analysis 1: Comparison: Placebo + Pioglitazone vs Linagliptin + Pioglitazone; Linagliptin vs. Placebo The odds-ratio is based on a logistic regression model including baseline HbA1c and previous antidiabetes medication; Test type: Superiority or Other; p = 0.0051, Regression, Logistic; Odds Ratio (OR) = 2.103, 95% CI [1.25 to 3.539]

10. Secondary Outcome: Percentage of Patients With HbA1c<7.0 at Week 24
Description: The percentage of patients with an HbA1c value below 7% at week 24 was calculated for each treatment arm. If a patient did not have an HbA1c value at week 24 they were considered a failure, so HbA1c above 7%.
Time Frame: Baseline and Week 24
Population: This population includes the Full Analysis Set (FAS). Non-completers were considered as failure imputation (NCF).
Measure: Number; unit: percentage of patients
Arm/Group | Placebo + Pioglitazone | Linagliptin + Pioglitazone
Number analyzed (Participants) | 128 | 252
percentage of patients | 30.5 | 42.9

11. Secondary Outcome: Percentage of Patients With HbA1c <6.5% at Week 24
Description: The percentage of patients with an HbA1c value below 6.5% at week 24 was calculated for each treatment arm. If a patient did not have an HbA1c value at week 24 they were considered a failure, so HbA1c above 6.5%. Only patients with baseline HbA1c >= 6.5%
Time Frame: Baseline and Week 24
Population: This population includes the FAS with baseline HbA1c >= 6.5%. Non-completers were considered as failure imputation (NCF).
Measure: Number; unit: percentage of patients
Arm/Group | Placebo + Pioglitazone | Linagliptin + Pioglitazone
Number analyzed (Participants) | 128 | 252
percentage of patients | 14.1 (0) | 17.5 (0)
Statistical Analysis 1: Comparison: Placebo + Pioglitazone vs Linagliptin + Pioglitazone; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.3547, Regression, Logistic; Odds Ratio (OR) = 1.348, 95% CI [0.716 to 2.537]

12. Secondary Outcome: Percentage of Patients With HbA1c<6.5% at Week 24
Description: The percentage of patients with an HbA1c value below 6.5% at week 24 was calculated for each treatment arm. If a patient did not have an HbA1c value at week 24 they were considered a failure, so HbA1c above 6.5%
Time Frame: Baseline and week 24
Population: This population includes the Full Analysis Set (FAS). Non-completers were considered as failure imputation (NCF).
Measure: Number; unit: percentage of patients
Arm/Group | Placebo + Pioglitazone | Linagliptin + Pioglitazone
Number analyzed (Participants) | 128 | 252
percentage of patients | 14.1 | 17.5

13. Secondary Outcome: Percentage of Patients Who Have an HbA1c Lowering by 0.5% at Week 24
Description: The percentage of patients with an HbA1c reduction from baseline greater than 0.5% at week 24 was calculated for each treatment arm. If a patient did not have an HbA1c value at week 24 they were considered a failure, so HbA1c reduction less than 0.5%.
Time Frame: Baseline and Week 24
Population: The Full Analysis Set (FAS) included all patients with a baseline and at least one on treatment HbA1c measurement available. Non-completers were considered as failure imputation (NCF).
Measure: Number; unit: percentage of patients
Arm/Group | Placebo + Pioglitazone | Linagliptin + Pioglitazone
Number analyzed (Participants) | 128 | 252
percentage of patients | 50.8 (0) | 75.0 (0)
Statistical Analysis 1: Comparison: Placebo + Pioglitazone vs Linagliptin + Pioglitazone; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 3.823, 95% CI [2.286 to 6.394]

ADVERSE EVENTS:
Time Frame: From day of first dose until 7 days after last dose, up to 202 days
Arm/Group | Placebo + Pioglitazone | Linagliptin + Pioglitazone
Serious Adverse Events (participants affected / at risk) | 3/130 | 8/259
Other Adverse Events (participants affected / at risk) | 21/130 | 33/259
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Pioglitazone (N=130) | Linagliptin + Pioglitazone (N=259)
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Glaucoma (Eye disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Meniscus removal (Surgical and medical procedures) | 0 | 1
Varicose vein (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Pioglitazone (N=130) | Linagliptin + Pioglitazone (N=259)
Nasopharyngitis (Infections and infestations) | 11 | 24
Upper respiratory tract infection (Infections and infestations) | 10 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.